CLINICAL TRIAL: NCT05444166
Title: Explore the Relationship Between the Percentage of Colonoscopy Withdrawal Overspeed and the Adenoma Detection Rate: a Prospective, Multicenter, Observational Study
Brief Title: Explore the Relationship Between the Percentage of Colonoscopy Withdrawal Overspeed and the ADR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Renmin Hospital of Wuhan University (Other)
Responsible Party: Sponsor
Other Study IDs: EA-22-020
Record Dates: First submitted 2022-06-29; First posted 2022-07-05 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Colonoscopy; Artificial Intelligence; Gastrointestinal Disease; Deep Learning
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Patient colonoscopy videos, photo documentation and pathological section
Oversight: FDA-regulated Drug: No

SUMMARY:
In this study, the investigators used the optical flow method to measure the colonoscopy withdrawal speed, and doctors were selected from multiple hospitals to collect prospective colonoscopy screening videos, and the percentage of colonoscopy withdrawal overspeed was calculated to explore the relationship between it based on optical flow method and the adenoma detection rate.

DETAILED DESCRIPTION:
Study showed that adequate withdrawal time is an important prerequisite for full mucosal inspection. In a large population-based analysis, a 1-min increase in withdrawal time led to a 3.6% increase in the ADR. Protocols or expert consensus recommend a standard withdrawal time of 6 min or longer. However, Findings of studies showed that a number of colonoscopies had a withdrawal time less than 6 min, which greatly reduces the ADR.

Investigator's preliminary experiments have shown that deep learning can monitor the colonoscopy withdrawal time in real-time and improve the adenoma detection rate. Based on the above rich foundation of preliminary work and the massive demand for improving the colonoscopy withdrawal assessment system.

The investigators improved EndoAngel to use optical flow method to monitor the colonoscopy withdrawal speed. The performance of the EndoAngel system was verified in colonoscopy videos. The investigators then aimed to evaluate whether the EndoAngel system could improve polyp detection rate after restricting the colonoscopy withdrawal speed.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years old;
2. Able to read, understand and sign an informed consent;
3. The investigator believes that the subjects can understand the process of the clinical study, are willing and able to complete all study procedures and follow-up visits, and cooperate with the study procedures;
4. Patients requiring screening colonoscopy.

Exclusion Criteria:

1. Have drug or alcohol abuse or mental disorder in the last 5 years;
2. Pregnant or lactating women;
3. Patients with known multiple polyp syndrome;
4. patients with known inflammatory bowel disease;
5. known intestinal stenosis or space-occupying tumor;
6. known colon obstruction or perforation;
7. patients with a history of colorectal surgery;
8. Patients with a previous history of allergy to pre-used spasmolysis;
9. Unable to perform biopsy and polyp removal due to coagulation disorders or oral anticoagulants;
10. High-risk diseases or other special conditions that the investigator considers the subject unsuitable for participation in the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this study, endoscopists who completed at least 140 colonoscopies were selected as the research objects, and patients who met the criteria were included in the experiment.
Sampling Method: Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2022-07-29 (Actual); Primary Completion 2023-10-29 (Estimated); Study Completion 2023-11-29 (Estimated)

PRIMARY OUTCOMES:
The adenoma detection rate (ADR) | A month
  ADR was calculated by dividing the total number of patients being detected adenomas by the number of colonoscopies.
The percentage of colonoscopy withdrawal overspeed | A month
  The percentage of colonoscopy withdrawal overspeed was calculated by dividing the time of colonoscopy withdrawal overspeed by the total time of colonoscopy withdrawal.

SECONDARY OUTCOMES:
The polyp detection rate (PDR) | A month
  PDR was calculated by dividing the total number of patients being detected polyps by the number of colonoscopies.
The mean number of polyps per patient (MNP) | A month
  MNP was calculated by dividing the total number of polyps by the number of colonoscopies.
The mean number of adenomas per patient (MAP) | A month
  MAP was calculated by dividing the total number of adenomas by the number of colonoscopies.
colonoscopy withdrawal time | A month
  The time is taken to finish the examination from the beginning of the ileocecal region.
colonoscopy forward time | A month
  The time is taken to go from the rectum to the ileocecal region.

CONTACTS AND LOCATIONS:
Locations (1):
- Renmin Hospital, Hubei, Wuhan, Hubei, China